CLINICAL TRIAL: NCT02735928
Title: Feasibility, Efficacy and Safety of Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) With Cisplatin in Women With Recurrent Ovarian Cancer: an Open-label, Single-arm Phase I-II Clinical Trial
Brief Title: Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Applied to Platinum-Resistant Recurrence of Ovarian Tumor
Acronym: PARROT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PARROT
Record Dates: First submitted 2016-02-08; First posted 2016-04-13 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Ovarian Epithelial Cancer Recurrent; Platinum-resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PIPAC (Experimental): PIPAC stands for Pressurized IntraPeritoneal Aerosol Chemotherapies. Enrolled patients will undergo to explorative laparoscopy as usual and PC index will be determined according to Fagotti score (PIV). Pathological response will be determined by serial peritoneal biopsies. Then a pressurized aerosol containing cisplatin followed by doxorubicin will be applied via a nebulizer. The PIPAC procedure can be repeated after 4-6 weeks until progression or limiting toxicity
  Interventions: Device: Pressurized intraperitoneal aerosol chemotherapy with cisplatin and doxorubicin

INTERVENTIONS:
Device: Pressurized intraperitoneal aerosol chemotherapy with cisplatin and doxorubicin — After insufflation of a 12 mmHg of capnoperitoneum at 37 °C, two balloon trocars will be placed. Parietal biopsies will be taken and ascites (< 500cc) will be removed. A nebulizer will be connected to a high-pressure injector and will be inserted into the abdomen through a trocar. A pressurized aerosol containing cisplatin at a dose of 10.5 mg/m2 body surface in 150 ml NaCl 0.9 % followed by doxorubicin at a dose of 2.1 mg/m2 body surface in a 50 ml NaCl 0.9% solution will be applied via a nebulizer immediately. Then, the system will be kept in steady-state for 30 min (i.e.: application time).
  Other Names: PIPAC

SUMMARY:
Patients with first recurrent resistance ovarian cancer and disease progression with peritoneal carcinomatosis will undergo PIPAC procedure. The primary end point is to determine the clinical benefit rate (CBR) of a pressurized intraperitoneal aerosol chemotherapy with a combination of cisplatin and doxorubicin.

DETAILED DESCRIPTION:
This study aims to investigate the therapeutic efficacy of PIPAC using cisplatin and doxorubicin in women with first recurrent resistance ovarian cancer and disease progression with peritoneal carcinomatosis. The primary objective of this study is to determine the Clinical Benefit Rate (CBR) according to RECIST/GCOG criteria after three cycles of PIPAC with PIPAC cisplatin and doxorubicin

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by first or second platinum resistant epithelial ovarian tumor recurrence.
* ECOG-performance status ≤ 3.
* Adequate respiratory, hepatic, cardiac, kidney and bone marrow function (absolute neutrophil count > 1500 / mm3, platelets > 150 000/μl, creatinine clearance > 60 mL / min according to Cockroft formula).
* Patient-compliant and psychologically able to follow the trial procedures.

Exclusion Criteria:

* Non-epithelial ovarian cancer or borderline ovarian tumor.
* Pregnancy or breastfeeding.
* Patients affected by major depressive disorder even in treatment or minor mood disorders.
* Patients with severe impairment of respiratory, hepatic or renal function.
* Patients with cardiac, neurological or metabolic uncontrolled pharmacologically disease
* Patients with bowel obstruction.
* Inadequate bone marrow, liver, kidney function.
* No clear-peritoneal disease at surgical exploration.
* Patients with ascites >2000 cc (CT-Scan)
* Patients who have already made third line chemotherapy.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit Rate (CBR) according to RECIST/GCOG criteria after three cycles of PIPAC with PIPAC cisplatin and doxorubicin | 12-18 weeks
  Evaluation of target lesions will be done as follows:
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  * Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase

SECONDARY OUTCOMES:
The median time to progression according to RECIST criteria after three cycles of PIPAC with cisplatin | 1 Year
  From the last chemotherapy cycle to the first clinical-radiological signs of disease relapse
Fagotti score, as assessed by laparoscopy | 1 Year
The degree of histological regression assessed by pathological review of repeated peritoneal biopsies | 1 Year
The proportion of women with a reduction of serum CA-125 of at least 50% after PIPAC | 1 Year
Evaluation of the Quality Of Life (QOL) on the basis of the European Organization for Research and Treatment of Cancer (EORTC) QOL questionnaires | 1 year
  Quality of life will be assess using the EORTC quality of life questionnaire core-36 (QLQC-30) and the ovarian cancer-specific quality of life questionnaire (QLQ-Ov28).These will be complete before and after the first, second, and third PIPAC applications

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fagotti A, Petrillo M, Costantini B, Fanfani F, Gallotta V, Chiantera V, Turco LC, Bottoni C, Scambia G. Minimally invasive secondary cytoreduction plus HIPEC for recurrent ovarian cancer: a case series. Gynecol Oncol. 2014 Feb;132(2):303-6. doi: 10.1016/j.ygyno.2013.12.028. Epub 2013 Dec 27. PMID 24378877
- [Result] Tempfer CB, Winnekendonk G, Solass W, Horvat R, Giger-Pabst U, Zieren J, Rezniczek GA, Reymond MA. Pressurized intraperitoneal aerosol chemotherapy in women with recurrent ovarian cancer: A phase 2 study. Gynecol Oncol. 2015 May;137(2):223-8. doi: 10.1016/j.ygyno.2015.02.009. Epub 2015 Feb 18. PMID 25701703
- [Result] Vizzielli G, Costantini B, Tortorella L, Petrillo M, Fanfani F, Chiantera V, Ercoli A, Iodice R, Scambia G, Fagotti A. Influence of intraperitoneal dissemination assessed by laparoscopy on prognosis of advanced ovarian cancer: an exploratory analysis of a single-institution experience. Ann Surg Oncol. 2014 Nov;21(12):3970-7. doi: 10.1245/s10434-014-3783-6. Epub 2014 May 22. PMID 24849521